CLINICAL TRIAL: NCT05082610
Title: A Phase 1 Study of HMBD-002-V4C26 (HMBD-002), a Monoclonal Antibody Targeting VISTA, as Monotherapy and Combined With Pembrolizumab, in Patients With Advanced Solid Malignancies
Brief Title: A Study of HMBD-002, a Monoclonal Antibody Targeting VISTA, as Monotherapy and Combined With Pembrolizumab, in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hummingbird Bioscience (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMBD-002-V4C26-01
Record Dates: First submitted 2021-09-21; First posted 2021-10-19 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Tumor, Solid; Nonsmall Cell Lung Cancer; Triple Negative Breast Cancer; Malignant Neoplasm; Metastatic Cancer; Advanced Solid Tumor
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 - Dose Escalation Phase (Monotherapy) (Experimental): HMBD-002 administered as a 60-minute IV infusion as a monotherapy. HMBD-002 will be administered on Days 1, 8, and 15 of a 21-day cycle.
  Interventions: Drug: HMBD-002
- Part 1 - Dose Escalation Phase (Combination Therapy) (Experimental): HMBD-002 administered as a 60-minute IV infusion at escalating doses in combination with pembrolizumab KEYTRUDA®. HMBD-002 will be administered on Days 1, 8, and 15 of a 21-day cycle.
  The treatment pembrolizumab KEYTRUDA® will be administered as a 30-minute IV infusion at a dose of 200 mg on Day 1 of every 21-day cycle.
  Interventions: Drug: HMBD-002; Drug: Pembrolizumab
- Part 2 - Dose Expansion (Monotherapy) (Experimental): HMBD-002 administered at the MTD/RP2D as a 60-minute IV infusion as a monotherapy in patients with TNBC or NSCLC.
  Interventions: Drug: HMBD-002
- Part 2 - Dose Expansion (Combination Therapy) (Experimental): HMBD-002 administered at the MTD/RP2D as a 60-minute IV infusion in combination with pembrolizumab KEYTRUDA® at the standard labeled dose in patients with TNBC or NSCLC.
  Interventions: Drug: HMBD-002; Drug: Pembrolizumab

INTERVENTIONS:
Drug: HMBD-002 — IgG4 monoclonal antibody (mAb) targeting the V-domain immunoglobulin suppressor of T cell activation (VISTA) receptor.
Drug: Pembrolizumab — IgG4 mAb with high specificity of binding to the PD-1 receptor, thus inhibiting its interaction with PD-L1 and programmed cell death ligand 2 (PD-L2).
  Arms: Part 1 - Dose Escalation Phase (Combination Therapy); Part 2 - Dose Expansion (Combination Therapy)

SUMMARY:
This is a phase 1/2, open-label, multi-center, first-in-human, two-stage (Part 1: dose escalation and Part 2: dose expansion) study evaluating multiple doses and schedules of intravenously (IV) administered HMBD-002, with or without pembrolizumab KEYTRUDA®, in patients with advanced solid tumors (i.e., locally advanced and unresectable, or metastatic).

DETAILED DESCRIPTION:
This is a phase 1/2, open-label, multi-center study whose principal phase 1 stage objective is to determine the recommended phase 2 dose (RP2D) of the anti-VISTA monoclonal antibody (mAb) as a single agent and combined with the anti-PD-1 mAb pembrolizumab KEYTRUDA® in subjects with advanced solid malignancies.

In the phase 2 stage, the antitumor activity of HMBD-002 alone or combined with pembrolizumab KEYTRUDA® will be evaluated in patients with triple negative breast cancer (TNBC), non-small cell lung cancer (NSCLC) and a wide range of other malignancies known or documented to express VISTA.

ELIGIBILITY:
Inclusion Criteria (Phase 1 and 2 Stages)

1. Histologic or cytologic evidence of a malignant solid cancer (any histology) with advanced or metastatic disease and no available therapies known to confer clinical benefit.
2. Tumor tissue, or paraffin block, ideally from the patient's most recent biopsy. A fresh tumor biopsy will be obtained if archival samples are not available.
3. Measurable by Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
4. At least 18 years old.
5. An Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
6. Adequate hematopoietic, kidney, and liver functions.
7. A left ventricular ejection fraction (LVEF) ≥ 45%.
8. Women of childbearing potential (WOCBP) must not be pregnant or breastfeeding. A WOCBP must agree to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
9. Male subjects must agree to follow contraceptive guidance during the study period and for at least 120 days after the last dose of study treatment.
10. Patient must give informed written consent for the study.

Inclusion Criteria for HMBD-002 Phase 2 Stage

Triple Negative Breast Cancer (TNBC)

1. Histologic or cytologic evidence of TNBC that is advanced or metastatic.
2. Will be requested to undergo a tumor biopsy before treatment and after 6 weeks of treatment.
3. Must have received appropriate treatment with at least one prior regimen for TNBC and there are no available therapies known to confer clinical benefit.

Non-Small Cell Lung Cancer (Monotherapy and Combination)

1. Histologic or cytologic evidence of NSCLC that is advanced or metastatic.
2. Will be requested to undergo a tumor biopsy before treatment and after 6 weeks of treatment.
3. Absence of an activating mutation of the EGFR or ALK.
4. Must have received treatment with an approved therapy if there are other genomic aberrations for which targeted therapies are approved and available.
5. Must have had disease progression on at least one approved or comparable standard therapy for NSCLC.
6. Must have received appropriate prior treatment with a mAb to PD-1 or PD-L1.

Multiple Other Cancers (Combination Therapy Baskets)

1. Histologic or cytologic evidence of an advanced or metastatic cancer aside from TNBC and NSCLC with no available therapies known to confer clinical benefit.
2. Will be requested to undergo a tumor biopsy before treatment and after 6 weeks of treatment.
3. Must have had appropriate treatment for their specific cancer and there is an absence of available therapy with a reasonable likelihood of conferring clinical benefit.

Exclusion Criteria

1. If the patient received prior therapy with an anti-PD-1 or anti-PD-L1 mAb or with an agent targeting stimulatory or co-inhibitory T-cell receptor and was discontinued from that treatment due to a Grade 3 or higher immune related adverse event.
2. Received radiotherapy within 2 weeks of treatment.
3. Received radiotherapy exceeding 30 Gray (Gy) to the lung within 6 months of the first dose of study medication.
4. Received an allogeneic tissue/solid organ transplant.
5. Received a live or live-attenuated vaccine within 30 days prior to the first dose of study medication.
6. Received a VISTA targeting agent.
7. The patient must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline.
8. The patient has an active autoimmune disease that required systemic treatment in the past.
9. Presence of an uncontrolled endocrine disorder.
10. Presence of clinically significant cardiovascular disease.
11. History of (non-infectious) pneumonitis or interstitial pulmonary disease that required steroids or has current pneumonitis or interstitial pulmonary disease.
12. Presence of uncontrolled, clinically significant pulmonary disease.
13. A previous a severe hypersensitivity reaction (≥ Grade 3) to pembrolizumab and/or any of its excipients.
14. A diagnosis of immunodeficiency or is receiving chronic systemic corticosteroids at a dose that exceeds 10 mg daily of prednisone equivalent or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
15. An uncontrolled intercurrent illness that would limit compliance with the study.
16. A positive status for human immunodeficiency virus (HIV).
17. A known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C viral (defined as HCV RNA detected) infection.
18. Oxygen-dependence.
19. A medical condition which, in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicity.
20. A positive COVID test within one week of study treatment if not fully vaccinated.
21. Another active malignancy that is progressing or has required active treatment within the past 3 years.
22. Known active central nervous system metastases and/or carcinomatous meningitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | First 21 days of treatment.
  The incidence of DLTs during the DLT assessment period.
Dose-Finding | Screening to 90 days from last dose.
  Determination of the MTD or maximum tested dose, and the RP2D.
Frequency and Severity of Adverse Events (AE) | Screening to 90 days from last dose.
  The incidences and percentages of patients experiencing AEs summarized by NCI CTCAE version 5.0 grade and by causality.

SECONDARY OUTCOMES:
Pharmacokinetics of HMBD-002 | Day 1 of dosing through 21 days post last dose.
  Maximum Plasma Concentration (Cmax)
Pharmacokinetics of HMBD-002 | Day 1 of dosing through 21 days post last dose.
  Area Under the Curve (AUC)
Objective Response Rate (ORR) | Day 1 of dosing through every 90 after the last dose.
  ORR according to RECIST v1.1.
Duration of Response (DoR) | Day 1 of dosing through every 90 after the last dose.
  Time from the date measurement criteria are first met for PR or CR to the date measurement criteria are first met for PD.
Progression Free Survival (PFS) | Day 1 of dosing through every 90 after the last dose.
  Time from the date of initiation of study therapy to the date measurement criteria are first met for PD or death from any cause, whichever occurs first.
Overall Survival (OS) | Day 1 of dosing through every 90 after the last dose.
  Time from the date of initiation of study therapy to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The City of Hope National Medical Center, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Smilow Cancer Hospital - Yale New Heaven Health, New Haven, Connecticut
  - UTSW Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No